CLINICAL TRIAL: NCT00310284
Title: Computerized Self-Help Treatment for Primary Insomnia
Brief Title: A Treatment Study Comparing Two Non-Drug, Self-Help Treatment of Chronic Insomnia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PICS, Inc. (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R44HL065893 (NIH); 5R44HL065893 (NIH)
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2006-03

CONDITIONS: Insomnia
Keywords: Insomnia; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

INTERVENTIONS:
Behavioral: Computerized delivery of cognitive-behavioral treatment of insomnia
Behavioral: Self-help manual to improve insomnia symptoms

SUMMARY:
The purpose of this study is to determine whether a handheld computer is superior to a self-help manual for the treatment of chronic primary insomnia.

DETAILED DESCRIPTION:
Chronic primary insomnia is a highly prevalent condition, affecting up to 15% of the population. The condition is associated with daytime fatigue, lack of concentration, and decreased quality of life. Most people with chronic primary insomnia go untreated, because of a desire to avoid medication or lack of access to quality non-drug treatments. Therefore, an affordable, easy to use, and effective computer to help assess and treat insomnia symptoms could bring treatment to this population.

Comparison: We are comparing a new handheld computer that uses cognitive-behavioral treatment principles to a popular self-help manual for the treatment of primary insomnia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* sleep less than 6.5 hours per night
* at least 30 minutes of sleep onset latency or wakefulness after sleep onset
* symptoms present for at least 6 months
* must have insomnia symptoms at least 3 days per week

Exclusion Criteria:

* Body Mass Index greater than 32
* Presence of anxiety disorder
* Secondary forms of insomnia
* Presence of a substance use disorder
* Concurrent treatment for another mental disorder
* History of other sleep disorders, including: apnea, restless legs, periodic limb movement disorder, or narcolepsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-01

PRIMARY OUTCOMES:
Changes in sleep parameters via polysomnography
Changes in sleep parameters via self-reported sleep diary
Changes in symptom severity as measured by Insomnia Severity Index
Changes in symptom severity as measured by Pittsburgh Sleep Quality Index
Changes in symptom severity as measured by the Multi-dimensional Fatigue Inventory

SECONDARY OUTCOMES:
Changes in depression symptoms as measured by Beck Depression Inventory II
Changes in quality of life as measured by a qualitative instrument
Usability of the device as measured by a qualitative questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bradford W Applegate, Ph.D., Principal Investigator — PICS, Inc.
Locations (1):
- PICS, Inc., Reston, Virginia, United States